CLINICAL TRIAL: NCT00126685
Title: Vaccination of Stage IV Cutaneous Melanoma Patients With Mature, Autologous Monocyte-Derived Dendritic Cells Transfected With Unselected Autologous Amplified Tumor-RNA
Brief Title: Vaccine Therapy in Treating Patients With Stage IV Melanoma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Dermatologische Klinik MIT Poliklinik-Universitaetsklinikum Erlangen (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000435933; ERLANGEN-DERMA-ER-DC-07; EU-20513; ARGOS-ERLANGEN-DERMA-DC-07
Record Dates: First submitted 2005-08-03; First posted 2005-08-04 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2007-06

CONDITIONS: Melanoma (Skin)
Keywords: stage IV melanoma; recurrent melanoma
MeSH Terms: conditions — Melanoma | interventions — FANG vaccine

INTERVENTIONS:
Biological: autologous tumor cell vaccine
Biological: therapeutic autologous dendritic cells

SUMMARY:
RATIONALE: Vaccines made from a person's tumor cells and white blood cells may help the body build an effective immune response to kill tumor cells.

PURPOSE: This phase I/II trial is studying the side effects of vaccine therapy and to see how well it works in treating patients with stage IV melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the safety and tolerability of vaccine therapy comprising autologous dendritic cells (DC) transfected with autologous polymerase chain reaction-amplified tumor RNA in patients with stage IV cutaneous melanoma.
* Determine whether tumor RNA- or tumor antigen-specific T-cell responses are induced in patients treated with this vaccine.
* Determine whether there are major differences in the immunogenicity of DC transfected at immature stage or at mature stage in patients treated with this vaccine.
* Determine objective tumor response in patients treated with this vaccine.
* Determine time to disease progression and progression-free interval in patients treated with this vaccine.
* Determine overall survival of patients treated with this vaccine.

OUTLINE: This is an open-label, nonrandomized study. Patients are sequentially assigned to receive dendritic cells (DC) transfected at either immature or mature stage.

Approximately 2-3 weeks before leukapheresis, patients undergo surgical excision or biopsy of the tumor to obtain tumor tissue for RNA isolation. RNA is amplified from the tumor sample by polymerase chain reaction (PCR). Patients then undergo leukapheresis to harvest peripheral blood mononuclear cells for the production of DC on day -14 . DC at immature or mature stage are transfected with autologous PCR-amplified tumor RNA to produce the vaccine. Patients receive vaccine intradermally (ID) on days 1, 15, 29, 43, 57, and between days 71-74 in the absence of disease progression or unacceptable toxicity. Patients undergo evaluation between days 71-74. Patients with responding or stable disease or minor disease progression receive booster vaccine ID on days 99, 127, between days 162-164, on day 205, between days 253-255, 351-354, 442-444, 533-535, 624-626, and 715-718 in the absence of disease progression or unacceptable toxicity. Patients also undergo additional leukapheresis between days 71-74, 351-354, and 715-718. Patients with responding or stable disease may continue to undergo leukapheresis and receive booster vaccine ID every 12-24 weeks off study.

After completion of study treatment, patients are followed periodically for up to 10 years.

PROJECTED ACCRUAL: A total of 8-30 patients will be accrued for this study within 6-12 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed cutaneous melanoma*

  * Stage IV disease (i.e., distant metastasis)
  * Not curable by surgical resection
* NOTE: *Metastatic melanoma with an unknown primary tumor allowed provided ocular melanoma can be definitely excluded and origin from the skin is likely
* Unidimensionally or bidimensionally measurable disease by physical examination and/or noninvasive radiological procedures

  * At least 1 measurable metastasis that has not been previously excised or biopsied
* Failed ≥ 1 standard chemotherapy or chemoimmunotherapy regimen (e.g., dacarbazine or cisplatin monotherapy)
* At least 1 metastatic lesion surgically accessible* for excision or biopsy to obtain tumor material for RNA isolation** NOTE: *Surgically accessible metastatic lesion not required provided properly processed tumor material or isolated tumor RNA is available from a metastasis excised or biopsied within the past 6 months

NOTE: **Major surgery not allowed for the acquisition of metastatic material solely for RNA isolation

* No active CNS metastases by CT scan or MRI

  * Previously treated CNS metastases (e.g., by excision of a single metastasis, gamma knife radiosurgery, or stereotactic radiotherapy) allowed provided there is no evidence of active CNS metastasis by CT scan or MRI

PATIENT CHARACTERISTICS:

Age

* Over 18

Performance status

* Karnofsky 60-100%

Life expectancy

* At least 4 months

Hematopoietic

* WBC > 2,500/mm^3
* Neutrophil count > 1,000/mm^3
* Lymphocyte count > 700/mm^3
* Platelet count > 75,000/mm^3
* Hemoglobin > 9 g/dL
* No bleeding disorders

Hepatic

* Bilirubin < 2.0 mg/dL
* Hepatitis B surface antigen negative
* Hepatitis C antibody negative

Renal

* Creatinine < 2.5 mg/dL

Cardiovascular

* No clinically significant heart disease

Pulmonary

* No respiratory disease

Immunologic

* HIV-1 or -2 negative
* Human T-cell lymphotropic virus type I negative
* No known hypersensitivity to dimethylsulfoxide
* No immunodeficiency disease
* No active systemic infection
* No active autoimmune disease (except vitiligo), including any of the following:

  * Lupus erythematosus
  * Scleroderma
  * Rheumatoid arthritis (i.e., rheumatoid factor-positive arthritis with current or recent flare)
  * Ankylosing spondylitis
  * Autoimmune thyroiditis or uveitis
  * Autoimmune hemolytic anemia
  * Immune thrombocytopenic purpura
  * Multiple sclerosis
  * Inflammatory bowel disease

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile female patients must use effective contraception during and for ≥ 4 weeks after completion of study treatment
* Willing to undergo excision or biopsy of metastasis
* Willing to be hospitalized for ≥ 24 hours after each vaccination
* Medical condition stable
* No contraindication to leukapheresis
* No organic brain syndrome
* No significant psychiatric abnormality that would preclude study participation
* No other active malignancy within the past 5 years except nonmelanoma skin cancer or carcinoma in situ of the cervix
* No other major serious illness

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Disease Characteristics
* More than 4 weeks since prior systemic immunotherapy
* No systemic immunotherapy during and for 2 weeks after completion of study treatment

Chemotherapy

* See Disease Characteristics
* More than 4 weeks since prior systemic chemotherapy
* No systemic chemotherapy during and for 2 weeks after completion of study treatment

Endocrine therapy

* No systemic corticosteroids, including steroid-containing inhalers or chronic use of topical steroids over large areas of the body (if systemic effects are likely or obvious) during and for 2 weeks after completion of study treatment

Radiotherapy

* See Disease Characteristics
* More than 2 weeks since prior radiotherapy
* No prior radiotherapy to the spleen
* Concurrent palliative radiotherapy to selected metastases for pain or local complications (e.g., compression) allowed

Surgery

* See Disease Characteristics
* Recovered from prior surgery
* No prior splenectomy
* No prior organ allograft
* Concurrent palliative surgery to selected metastases for pain or local complications (e.g., compression) allowed

Other

* Concurrent palliative hyperthermic therapy to selected metastases for pain or local complications (e.g., compression) allowed
* No concurrent participation in any other clinical trial
* No other systemic immunosuppressive agents (e.g., azathioprine or cyclosporine) during and for 2 weeks after completion of study treatment
* No other investigational drugs or paramedical substances during and for 2 weeks after completion of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2005-04

PRIMARY OUTCOMES:
Safety
Immunogenicity
Objective tumor response
Time to disease progression
Progression-free interval
Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Gerold Schuler, Study Chair — Dermatologische Klinik MIT Poliklinik-Universitaetsklinikum Erlangen
Locations (1):
- Dermatologische Klinik mit Poliklinik - Universitaetsklinikum Erlangen, Erlangen, Germany